CLINICAL TRIAL: NCT04818723
Title: Role of Montelukast in Preventing Relapse in Childhood Idiopathic Nephrotic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nishtar Medical University (Other)
Responsible Party: Principal Investigator, Hashim Raza, Principal Investigator, Nishtar Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NishtarMU
Record Dates: First submitted 2021-03-22; First posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Nephrotic Syndrome
Keywords: Leukotriene antagonists; Nephrotic syndrome; Steroid
MeSH Terms: conditions — Nephrotic Syndrome | interventions — montelukast

STUDY DESIGN:
Intervention Model Description: During the study period, adopting non-probability consecutive sampling method, patients were assigned into two groups; 53 in Case Group (given montelukast 5mg at bed time) and 53 in Control Group (given no montelukast).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Montelukast Group (Experimental): 53 in Case Group (given montelukast 5mg at bed time). All patients were induced with prednisolone 2mg/kg single morning dose with breakfast for total 4 weeks. Patients who did not achieve remission after 4 weeks' full dose were labeled steroid resistant nephrotic syndrome (SRNS). Children with steroid sensitive nephrotic syndrome SSNS were further treated by prednisolone 1.5 mg/kg single morning dose with breakfast every other day for the next 4 weeks. Prednisolone was then tapered by reducing 25% dose fortnightly and completely stopped in 8 weeks. Patients in the Case Group continued taking montelukast after stopping steroids. All patients were followed up every 4-8 weeks for a minimum of 12 months to look for response to treatment, side effects of medications, other co-morbidities, and the number of relapses. Relapses were treated with repeat prednisolone doses according to the protocol of treatment for relapse.
  Interventions: Drug: Montelukast
- Placebo Group (Placebo Comparator): Patients in this groups were induced with prednisolone 2mg/kg single morning dose with breakfast for total 4 weeks. Patients who did not achieve remission after 4 weeks' full dose were labeled steroid resistant nephrotic syndrome (SRNS). Children with steroid sensitive nephrotic syndrome SSNS were further treated by prednisolone 1.5 mg/kg single morning dose with breakfast every other day for the next 4 weeks. Prednisolone was then tapered by reducing 25% dose fortnightly and completely stopped in 8 weeks. Patients in the Case Group continued taking montelukast after stopping steroids. All patients were followed up every 4-8 weeks for a minimum of 12 months to look for response to treatment, side effects of medications, other co-morbidities, and the number of relapses. Relapses were treated with repeat prednisolone doses according to the protocol of treatment for relapse.
  Interventions: Drug: Montelukast

INTERVENTIONS:
Drug: Montelukast — We wanted to know the role of leukotriene receptor antagonist (LTRA) montelukast in preventing relapses in idiopathic childhood nephrotic syndrome (NS)

SUMMARY:
The investigators planned this research to elucidate if there is any efficacy of montelukast, a leukotriene receptor antagonist, in steroid sensitive childhood onset NS to help prevent relapses. This study was done to know the role of leukotriene receptor antagonist (LTRA) montelukast in preventing relapses in idiopathic childhood nephrotic syndrome (NS)

DETAILED DESCRIPTION:
A quasi-experimental study, done at Department of Pediatric Nephrology at the Children's Hospital & the Institute of Child Health, Multan. A total of 96 patients aged 1-10 years with steroid sensitive Idiopathic NS were assigned into two groups (48 patients in each group). The case group received montelukast 5mg daily at bed time while the control group was not given montelukast. Steroid treatment protocol was the same for the two groups as per institutional guidelines. Patients were monitored and followed for the response to treatment and evidence of relapse over the study period (minimum 12 months).

ELIGIBILITY:
Inclusion Criteria:A total of 106 children aged 1-10 years with idiopathic nephrotic syndrome were enrolled

-

Exclusion Criteria: - Patients having Steroid resistant nephrotic syndrome (SRNS) or those having nephrotic syndrome with atypical features or Secondary cause were excluded.

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Prevention of relapse in idiopathic childhood nephrotic syndrome | 1 year
  Relapse was labeled as recurrence of proteinuria 3+ or more for 3 consecutive days with or without edema

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatric Nephrology, The Children's Hospital and Institute of Child Health, Multan, PPunjab, Pakistan